CLINICAL TRIAL: NCT03596320
Title: Yield of Colonoscopy in Children With Bleeding Per Rectum Attending Gastrointestinal Endoscopic Unit In Assuit University Children Hospital
Brief Title: Yield of Colonoscopy in Children With Rectal Bleeding
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, SHIraqi, principle investigator, Assiut University
Other Study IDs: crbchildren
Record Dates: First submitted 2018-07-07; First posted 2018-07-23 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Colonic Diseases
MeSH Terms: conditions — Colonic Diseases | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: colonoscopy — description of the results of colonoscopy im managment of children with rectal bleeding

SUMMARY:
description study of colonscopy in children with bleeding per rectum attending gastrointestinal endoscopic unit in assiut university children hospital from 2014-2019

DETAILED DESCRIPTION:
Rectal bleeding is a source of anxiety for both children and parents and is frequently encountered clinical complaint in routine practice in pediatric patient . Lower gastrointestinal bleeding means bleeding from sites distal to the ligament of treitz and presents as rectal bleeding while passage of bright red blood from the rectum is called hematochezia.

The etiology of rectal bleeding is different in children than in adult according to age group which enables physicians to make appropriate differential diagnosis. There are several etiologies for rectal bleeding in pediatric practice ranging from mild condition requiring little or no treatment to severe and life-threating ones requiring immediate intervention. The etiologies include anal fissure, food allergy, infectious enterocolitis, Meckel'sdiverticulum, intussusceptions, volvulus, lymphonodular hyperplasia, inflammatory bowel disease, angiodysplasia, hemorrhoids, and hemolytic -uremic syndrome. Common causes of bleeding per rectum in children vary between studies . Once the bleeding is suspected to be coming from lower gastrointestinal tract it warrant an evaluation in all cases by proctosigmoidoscopy followed by colonoscopy .

Colonoscopy is the examination of choice for diagnosis and management of bleeding per rectum in children . The benefits of colonoscopy include identification of the site of bleeding regardless of the rate or presence of bleeding through visualization the entire length of the colon often include the distal ileum by possibility of endoscpic intervention and biopsy taking to make and confirm the diagnosis and follow up evaluation, so gastrointestinal endoscopy with biopsy is an essential tool for diagnosis of crohns disease and ulcerative colitis in children, as well as therapeutical intervention of colonoscopy by hemostasis, removing polyps, dilating stricture or decompressing the obstructed bowel .

Colonoscopy is considered a safe and low risk procedure. Complications of colonoscopy are rare and usually minor, as adverse effects of sedative medicine as (nausea,vomiting or allergies) can ocurr.

Bleeding after colonoscopy is usually minimal but may follow mucous biopsy or polypectomy, Perforation is very rare but it is the most serious complication of colonoscopy in children, it is usually related to polypectomy and can be successfully managed with surgical intervention. In case of infection in which cause the child will be given antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* all children with rectal bleeding underwent colonoscopy

Exclusion Criteria:

* children underwent colonoscopy rather than rectal bleeding

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: all children with bleeding per rectum underwent colonoscopy
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-07-20 (Estimated); Primary Completion 2019-05-30 (Estimated); Study Completion 2019-07-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants free and recurrance of colonic disease after colonoscopy procedure | 2 year
  Number of participants were monitored with recurrance of rectal bleeding and underwent colonoscopy up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Soha Iraqi, Principal Investigator — Assiut University
Locations (1):
- Assiut U, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GELB AM, MINKOWITZ S, TRESSER M. Rectal and colonic polyps occurring in young people. N Y State J Med. 1962 Feb 15;62:513-8. No abstract available. PMID 13897571
- [Background] Baxter NN, Goldwasser MA, Paszat LF, Saskin R, Urbach DR, Rabeneck L. Association of colonoscopy and death from colorectal cancer. Ann Intern Med. 2009 Jan 6;150(1):1-8. doi: 10.7326/0003-4819-150-1-200901060-00306. Epub 2008 Dec 15. PMID 19075198
- [Background] Bai Y, Peng J, Gao J, Zou DW, Li ZS. Epidemiology of lower gastrointestinal bleeding in China: single-center series and systematic analysis of Chinese literature with 53,951 patients. J Gastroenterol Hepatol. 2011 Apr;26(4):678-82. doi: 10.1111/j.1440-1746.2010.06586.x. PMID 21083610
- [Background] Fox VL. Gastrointestinal bleeding in infancy and childhood. Gastroenterol Clin North Am. 2000 Mar;29(1):37-66, v. doi: 10.1016/s0889-8553(05)70107-2. PMID 10752017
- [Result] Ladas SD, Karamanolis G, Ben-Soussan E. Colonic gas explosion during therapeutic colonoscopy with electrocautery. World J Gastroenterol. 2007 Oct 28;13(40):5295-8. doi: 10.3748/wjg.v13.i40.5295. PMID 17879396
- [Result] Park JH. Role of colonoscopy in the diagnosis and treatment of pediatric lower gastrointestinal disorders. Korean J Pediatr. 2010 Sep;53(9):824-9. doi: 10.3345/kjp.2010.53.9.824. Epub 2010 Sep 13. PMID 21189966
- [Result] Zahmatkeshan M, Fallahzadeh E, Najib K, Geramizadeh B, Haghighat M, Imanieh MH. Etiology of lower gastrointestinal bleeding in children:a single center experience from southern iran. Middle East J Dig Dis. 2012 Oct;4(4):216-23. PMID 24829660
- See also: Ting wu C, Chen C. Characteristics and diagnostic yield of pediatric colonoscopy in Taiwan, Pediatric of neonatology 2015; 56(5): 334-8 — https://doi.org/10.1016/j.pedneo.2015.01.005
- See also: Tringali A,Balassone V,Angelis P.Complication in pediatric colonoscopy.2015;30(5):825-39. — https://doi.org/10.1016/j.bpg.2016.09.006